CLINICAL TRIAL: NCT00292383
Title: A Randomized, Prospective Multicenter Pilot Study to Determine the Influence of the Ventricular Pacing Site on the Incidence of Atrial Fibrillation and Heart Failure in Patients With Indication for Permanent Pacemaker Stimulation Therapy.
Brief Title: Ventricular Pacing Site Selection (V-PASS)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medtronic BRC (Industry)
Collaborators: Vitatron GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V-PASS V.1.2.
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2007-10

CONDITIONS: Atrioventricular Block
Keywords: Cardiac Pacing, artificial; Atrial Fibrillation; Heart failure; Pacemaker leads; Lead position; Higher degree AV-Block
MeSH Terms: conditions — Atrioventricular Block; Atrial Fibrillation; Heart Failure

INTERVENTIONS:
Procedure: Leads to be implanted according randomization on specified sites. Vitatron pacemakers to be implanted: T60 DR, T70 DR, T20 SR, C60 DR

SUMMARY:
The purpose of this study is to determine whether there is a relationship between ventricular lead position and the incidence of heart failure and atrial fibrillation in patients with indication for permanent pacemaker stimulation.

DETAILED DESCRIPTION:
AV-Block of higher degree is the primary indication for pacing therapy for about 20% of pacemaker patients. Pacing systems with only ventricular stimulation (VVI and VDD) have a fraction of about 40% of all pacemakers in Germany. About 50% of the implanted pacemakers in Germany are dual-chamber pacemakers and one half of them is used for treatment of AV blocks.

Picture 1: Fractions of pacing indications in Germany Picture 2: Fractions of used pacing modes in Germany /1/

A lot of studies proved in the past that the pacing site influenced the development of hemodynamics, heart failure (HF) and atrial fibrillation (AF). Unfortunately, the results are not commonly applicable or statistically assured. Due to this, further examinations are required in order to get explicit statements regarding application of alternative, nonapical ventricular lead positioning.

1. Pilotphase It shall be determined whether a randomized positioning of ventricular leads at 2 defined positions (either Group A: Positioning at right ventricular apex or Group B:. Positioning at right ventricular high septum) is feasible. Included patients will already by examined and followed according to protocol. After having proved feasibility of randomized positioning, the data of these patients shall be used for evaluation of the V-PASS study.
2. Study Phase It shall be evaluated how far 2 defined different ventricular lead positions for permanent pacemaker therapy can influence the combined study endpoint mortality and clinically relevant symptoms of heart failure. Further more the development of hemodynamics and the incidence of atrial fibrillation shall be studied.

ELIGIBILITY:
Inclusion Criteria:

Patients with an expected ventricular stimulation rate of >60% in planned pacing therapy. This will be the following pacing indications

* Symptomatic first-degree AV block, PQ time >250ms
* Second-degree Av block with permanent 2:1 conduction
* Permanent third-degree AV block
* Paroxysmal first-degree to third-degree Av block, with an anticipated rate of ventricular stimulation >60%
* Symptomatic bradyarrhythmia absoluta with permanent atrial fibrillation, with an anticipated rate of ventricular stimulation >60%

Exclusion Criteria:

* heart failure acc. NYHA III or IV
* Intra-atrial conduction delay (P-wave > 150ms)
* Myocardial infarction less then 6 months before pacemaker implant
* hypertrophic obstructive cardiomyopathy
* Cardiogenic shock
* pregnancy
* Lactation period
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Study Completion 2008-12

PRIMARY OUTCOMES:
Amount of patients in which the ventricular lead position could be positioned successfully according randomization

SECONDARY OUTCOMES:
Typical values re operation procedure in both groups
operation time, x-ray time
intraoperative measurements (amplitudes, thresholds)
broad QRS-complexes in both groups
safety of therapy, complications
electrical specific values in both groups
energy consumption, lead impedance
Rhythmologic characteristics in both groups
amount of VESs
episodes of ventricular tachycardia
amount of atrial and ventricular stimulation
BNP-levels in both groups
incidence of co-morbidities in both groups
Atrial Fibrillation, AF burden >1%
Heart failure > NYHA II
Hospitalizations in both groups due to
Heart failure
Rhythm disorders

CONTACTS AND LOCATIONS:
Overall Officials: Jochem F. Stockinger, MD, Principal Investigator — Herzzentrum Bad Krozingen
Locations (3):
- Germany (3):
  - Herzzentrum Bad Krozingen, Elektrophysiologie, Bad Krozingen
  - Universitätsklinikum Heidelberg, Innere Medizin III, Heidelberg
  - Oberschwaben Klinik GmbH, Krankenhaus Wangen, Innere Med., Wangen

REFERENCES:
- [Background] Fachgruppe Herzschrittmacher. Bericht des Deutschen Herzschrittmacher Registers 2003 http://www.pacemaker-register.de/pdf/zentralregister_herzschrittmacher_bericht03.pdf
- [Background] DÄNISCHES HERZSCHRITTMACHERREGISTER http://www.pacemaker.dk
- [Background] SCHWEIZER HERZSCHRITTMACHERREGISTER http://www.pacemaker.ch
- [Background] Lemke B, Nowak B, Pfeiffer D; Deutschen Gesellschaft fur Kardiologie--Herz- und Kreislaufforschung e.V. Bearbeitet im Auftrag der Kommission fur Klinische Kardiologie. [Guidelines for heart pacemaker therapy]. Z Kardiol. 2005 Oct;94(10):704-20. doi: 10.1007/s00392-005-0269-3. No abstract available. German. PMID 16200488
- [Background] Gregoratos G., Abrams J. Epstein AE, et al. ACC/AHA /NASPE 2002 guideline update for implantation of cardiac pacemakers and antiarrhythmia devices: a report of the American College of Cardiology/ American Heart Association Task Force on Practice Guidelines (ACC/AHA/NASPE Committee on Pacemaker Implantation)(2002). http://www.acc.org/clinical/guidelines/pacemaker/pacemaker.pdf
- [Background] Lamas GA, Lee KL, Sweeney MO, Silverman R, Leon A, Yee R, Marinchak RA, Flaker G, Schron E, Orav EJ, Hellkamp AS, Greer S, McAnulty J, Ellenbogen K, Ehlert F, Freedman RA, Estes NA 3rd, Greenspon A, Goldman L; Mode Selection Trial in Sinus-Node Dysfunction. Ventricular pacing or dual-chamber pacing for sinus-node dysfunction. N Engl J Med. 2002 Jun 13;346(24):1854-62. doi: 10.1056/NEJMoa013040. PMID 12063369
- [Background] Frohlig G, Schwaab B, Kindermann M. Selective site pacing: the right ventricular approach. Pacing Clin Electrophysiol. 2004 Jun;27(6 Pt 2):855-61. doi: 10.1111/j.1540-8159.2004.00547.x. PMID 15189516
- [Background] Koglek W, Kranig W, Kowalski M, Kronski D, Brandl J, Oberbichler A, Suntinger A, Wutte M, Grimm G, Grove R, Ludorff G. [A simple method for AV-delay determination in dual chamber pacemakers]. Herzschrittmacherther Elektrophysiol. 2000 Dec;11(4):244-53. doi: 10.1007/s003990070023. German. PMID 27515355
- [Background] Giudici MC, Thornburg GA, Buck DL, Coyne EP, Walton MC, Paul DL, Sutton J. Comparison of right ventricular outflow tract and apical lead permanent pacing on cardiac output. Am J Cardiol. 1997 Jan 15;79(2):209-12. doi: 10.1016/s0002-9149(96)00718-7. PMID 9193029